CLINICAL TRIAL: NCT00830479
Title: A Randomized Trial of Endoscopic vs. Open Anti-Reflux Surgery For Treatment of Low-Grade Vesicoureteral Reflux: Surgical Treatment of Reflux: Endoscopic vs. Traditional CHoices (STRETCH) Study
Brief Title: Study of Endoscopic Versus Open Surgery for Urinary Reflux
Acronym: STRETCH
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to enroll patients for randomization
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Caleb Nelson, MD, MPH / PI, Children's Hospital Boston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-08-0354
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2011-08

CONDITIONS: Vesicoureteral Reflux
MeSH Terms: conditions — Vesico-Ureteral Reflux | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Open Surgery (Active Comparator)
  Interventions: Procedure: Anti-reflux surgery
- Endoscopic Surgery (Active Comparator)
  Interventions: Procedure: Endoscopic injection

INTERVENTIONS:
Procedure: Anti-reflux surgery — Open ureteroneocystostomy for correction of vesicoureteral reflux
  Arms: Open Surgery
Procedure: Endoscopic injection — Endoscopic injection of dextranomer/hyaluronic acid gel (Deflux) for correction of vesicoureteral reflux
  Arms: Endoscopic Surgery

SUMMARY:
This study seeks to compare outcomes after anti-reflux surgery (ARS) for correction of low-grade vesicoureteral reflux (VUR). It is a randomized controlled open-label trial of conventional open anti-reflux technique versus endoscopic anti-reflux technique with injection of dextranomer/hyaluronic acid copolymer (Deflux). Primary endpoint will be resolution of VUR at initial cystogram after ARS. Secondary outcomes will include incidence of postoperative UTI, resolution of VUR at 1-year cystogram after ARS, surgical complications, and quality of life measures after ARS.

ELIGIBILITY:
Inclusion Criteria:

* Age <12 years
* Unilateral or Bilateral Primary VUR
* Grade 2 or 3 (VCUG) or Grade 2 (RNC) VUR in at least 1 ureter
* Recommended for surgical correction of VUR by Urologist

Exclusion Criteria:

* Grade 4 or 5 (VCUG) or Grade 3 (RNC) VUR
* Secondary VUR (neurogenic bladder, exstrophy, or other causes of secondary VUR)
* Ureterocele
* Periureteral diverticulum
* Complete duplication of duplex collecting system on side with VUR
* Prior ARS, either open or endoscopic, regardless of success or failure
* History of other prior urinary tract surgery other than circumcision
* Solitary functional kidney
* Congenital or acquired immunodeficiency
* Chronic renal insufficiency or renal failure

Max Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Resolution of VUR at 4 months | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States